CLINICAL TRIAL: NCT03579381
Title: Specimen Repository for HIV Immunopathogenesis
Status: Completed | Type: Observational
Sponsor: AIDS Healthcare Foundation (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: AHF 03
Record Dates: First submitted 2018-01-09; First posted 2018-07-06 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: HIV-1-infection; Acute HIV Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMCs and Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immune Controllers: Patients with very low or undetectable levels of viremia without treatment
- Acute Infection: Early infection, i.e. within 2 weeks of infection

SUMMARY:
Specimen Repository for HIV Immunopathogenesis Studies

DETAILED DESCRIPTION:
The goal is to build a large specimen repository for collaborating scientists to run studies of immunity and HIV-1.

ELIGIBILITY:
Inclusion Criteria:

1. HIV positive (acutely infected, viremic and elite controllers)
2. Signed Informed Consent Form
3. Age at least 18 years old
4. Immune controllers, two types: "Elite suppressors" (HIV-positive with any three consecutive plasma HIV-1 RNA PCR undetectable while off treatment) or "viremic suppressors" (HIV-positive with any three consecutive HIV-1 RNA PCR <3000 while off treatment).
5. Acutely infected subjects:

Persons identified to have a negative HIV antibody response (ELISA) but positive detection of HIV-1 in the blood (RT-PCR) or individuals who have evidence of a recent (past 30 days) HIV negative result along with a current HIV positive result.

Exclusion Criteria:

1. Uncontrolled bleeding diathesis.
2. Pregnant.
3. Inability to provide informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acutely HIV infected individuals HIV infected individuals who are not on anti-retrovirals and have a viral load between 50 and 3,000 HIV infected individuals who are not on anti-retrovirals and have a viral load less than 49
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
HIV progression from acute infection to viral suppression | 2 years
  Outcomes will depend on scientists who use the samples for further study
HIV progression and control by elite and viremic suppressors | 2 years
  Outcomes will depend on scientists who use the samples for study

CONTACTS AND LOCATIONS:
Overall Officials: Otto O Yang, MD, Study Director — Scientific Director
Locations (1):
- AIDS Healthcare Foundation - Public Health Division, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No